CLINICAL TRIAL: NCT02996032
Title: CRUSH STUDY: Calculating Readmission Risk by Ultrasound for Heart Failure Study
Brief Title: CRUSH STUDY: Calculating Readmission Risk by Ultrasound for Heart Failure Failure Study
Acronym: CRUSH
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: Heart Failure Society of America (Unknown); Emergency Medicine Foundation (Other)
Responsible Party: Principal Investigator, Joseph Pare, Assistant Professor of Emergency Medicine, Boston Medical Center
Other Study IDs: H-35112
Record Dates: First submitted 2016-11-30; First posted 2016-12-19 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Heart Failure: Patients admitted to the hospital with acute decompensated heart failure expected to be hospitalized for at least 72 hours
  Interventions: Other: Vascular and Pulmonary Ultrasound

INTERVENTIONS:
Other: Vascular and Pulmonary Ultrasound

SUMMARY:
This is a study to determine if two ultrasound measures (Corrected Flow Time and B-Lines) can predict patients at higher risk of readmission within 30 days of hospital discharge for decompensated heart failure.

DETAILED DESCRIPTION:
Heart failure (HF) resulting in congestion is the leading cause for admission in persons ≥65 years of age and 20-25% of such patients are readmitted within 30 days of discharge. Efforts to treat HF are difficult without a simple method to detect early signs of congestion to direct therapy. Ultrasound can detect evidence of congestion by increased cardiac filling pressures two weeks prior to other markers of congestion such as weight gain or patient symptoms. Corrected flow time (FTc) measured by ultrasound, is an easy to perform vascular measure and correlates with cardiac filling pressures. Despite the relationship between FTc and filling pressures, this measure has never been studied in HF. The primary aim is to determine if FTc can predict patients at risk of readmission within 30 days. As a secondary aim, the investigators plan to validate a small study of patients reporting the ability of pulmonary ultrasound to predict readmissions. This study demonstrated pulmonary ultrasound was 100% sensitive and 68% specific for predicting readmission at 3 months, however this investigation was small and validation is needed. It is expected ultrasound will be able to accurately and safely predict patients who will be readmitted within 30 days of discharge. This proposal is aimed at identifying a noninvasive measure to better assess congestion from HF and predict readmissions.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Being admitted for heart failure with expected hospital stay of 72 hours

Exclusion Criteria:

* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with a diagnosis of acute decompensated heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in Corrected Flow Time | Measured daily during hospitalization and then correlated to 30 day readmissions.Mean hospitalization for the study population is 9 days, but will be measured during the duration of their hospitalization.
  Daily corrected flow time measures will be obtained during hospitalization. Mean hospitalization time for the study population is 9 days, but will be measured during the duration of their hospitalization. Changes in corrected flow time values will be assessed for associations with 30 day return visits. 30 Day returns will be determined by medical record review as well as follow up phone calls to patients. Corrected Flow Time is a single measure performed serial with the same units of measure.

SECONDARY OUTCOMES:
Change in Pulmonary Ultrasound (B-Lines) | Measured daily during hospitalization and correlated to 30 day readmissions. Mean hospitalization time for the study population is 9 days, but will be measured during the duration of hospitalization.
  Daily pulmonary ultrasound measures will be obtained during hospitalization. Mean hospitalization time for the study population is 9 days, but will be measured for the duration of their hospitalization. Changes in lung ultrasound values will be assessed for associations with 30 day return visits. 30 Day returns will be determined by medical record review as well as follow up phone calls to patients. Lung Ultrasound is a single measure performed serial with the same units of measure.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pare, MD MHS RDMS, Principal Investigator — Assistant Professor
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No